CLINICAL TRIAL: NCT03192215
Title: AtRial Cardiopathy and Antithrombotic Drugs In Prevention After Cryptogenic Stroke
Acronym: ARCADIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The DSMB halted the trial prematurely due to futility without any safety concerns.
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Cincinnati (Other); Medical University of South Carolina (Other); Bristol-Myers Squibb (Industry); Pfizer (Industry); Roche Pharma AG (Industry); Weill Medical College of Cornell University (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Randolph S. Marshall, MD, Elisabeth K Harris Professor of Neurology Chief, Stroke Division, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAR4607; 1U01NS095869-01A1 (NIH)
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Atrial Cardiopathy; Cryptogenic stroke; Ischemic stroke; Apixaban; Aspirin
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — apixaban; Aspirin

STUDY DESIGN:
Intervention Model Description: Active treatment will be either apixaban 5 mg or aspirin 81 mg. An adjusted dose of apixaban 2.5 mg will be used for subjects with at least two of the following: age greater than or equal to 80 years, body weight less than or equal to 60 kg, or known serum creatinine greater than or equal to 1.5 mg/dL. There will be six possible study tablets: apixaban 5 mg (regular dose), apixaban 2.5 mg (adjusted dose), apixaban 5 mg placebo, apixaban 2.5 mg placebo, aspirin 81 mg, and aspirin placebo.
  All subjects will be randomized to receive active treatment with either active apixaban or active aspirin. Study treatments will be supplied in a double-dummy fashion as apixaban 5 mg (2.5 mg for the adjusted dose) or matching placebo, and aspirin 81 mg or matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible patients will be allocated in a 1:1 ratio to apixaban or aspirin using the minimal sufficient balance randomization method to prevent serious treatment imbalances by study site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active agent: Apixaban (Experimental): Patients with a recent embolic stroke of undetermined source (ESUS) and evidence of atrial cardiopathy will receive Apixaban
  Interventions: Drug: Apixaban
- Active control: Aspirin (Active Comparator): Patients with a recent embolic stroke of undetermined source (ESUS) and evidence of atrial cardiopathy will receive Aspirin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Apixaban — 5 mg by mouth twice daily (2.5 mg for subjects meeting standard criteria for an adjusted dose).
  Other Names: Eliquis
  Arms: Active agent: Apixaban
Drug: Aspirin — Aspirin 81 mg by mouth once daily.
  Other Names: Aspirin Tablet
  Arms: Active control: Aspirin

SUMMARY:
Objectives

* Primary: To test the hypothesis that apixaban is superior to aspirin for the prevention of recurrent stroke in patients with cryptogenic ischemic stroke and atrial cardiopathy.
* Secondary: To test the hypothesis that the relative efficacy of apixaban over aspirin increases with the severity of atrial cardiopathy.

DETAILED DESCRIPTION:
ARCADIA is a multicenter, biomarker-driven, randomized, double-blind, active-control, phase 3 clinical trial of apixaban versus aspirin in patients who have evidence of atrial cardiopathy and a recent stroke of unknown cause. Eleven hundred subjects will be recruited over 2.5 years at up to 200 sites in and out of the NINDS StrokeNet consortium. Subjects will be followed for a minimum of 1.5 years and a maximum of 7 years for the primary efficacy outcome of recurrent stroke and the primary safety outcomes of symptomatic intracranial hemorrhage and major hemorrhage other than intracranial hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years.
* Clinical diagnosis of ischemic stroke + brain imaging to rule out hemorrhagic stroke.
* Modified Rankin Scale (MRS) score ≤ 4.
* Ability to be randomized within 3 to 180 days after stroke onset.
* ESUS, defined as all of the following:

  * Stroke detected by CT or MRI that is not lacunar. Lacunar is defined as a subcortical (this includes pons and midbrain) infarct in the distribution of the small, penetrating cerebral arteries whose largest dimension is ≤1.5 cm on CT or ≤2.0 cm on MRI diffusion images/<1.5 cm on T2 weighted MR images. The following are not considered lacunes: multiple simultaneous small deep infarcts, lateral medullary infarcts, and cerebellar infarcts. Patients with a clinical lacunar stroke syndrome and no infarct on imaging are excluded.
  * Absence of extracranial or intracranial atherosclerosis causing ≥50 percent luminal stenosis of the artery supplying the area of ischemia. Patients must undergo vascular imaging of the extracranial and intracranial vessels using either catheter angiography, CT angiogram (CTA), MR angiogram (MRA), or ultrasound, as considered appropriate by the treating physician and local principal investigator.
  * No major-risk cardioembolic source of embolism, including intracardiac thrombus, mechanical prosthetic cardiac valve, atrial myxoma or other cardiac tumors, moderate or severe mitral stenosis, myocardial infarction within the last 4 weeks, left ventricular ejection fraction <30 percent, valvular vegetations, or infective endocarditis). Patent foramen ovale is not an exclusion. All patients must undergo electrocardiogram, transthoracic or transesophageal echocardiography (TTE or TEE) and at least 24 hours of cardiac rhythm monitoring (Holter monitor or telemetry or equivalent). Additional cardiac imaging, such as cardiac MRI, or cardiac CT will be performed at the discretion of the local treating physician and principal investigator. Additional cardiac rhythm monitoring, such as monitored cardiac outpatient telemetry (MCOT) or an implanted cardiac monitor, will be at the discretion of the treating physician and local principal investigator.
  * No other specific cause of stroke identified, such as arteritis, dissection, migraine, vasospasm, drug abuse, or hypercoagulability. Special testing, such as toxicological screens, serological testing for syphilis, and tests for hypercoagulability, will be performed at the discretion of the treating physician and local principal investigator.

Exclusion Criteria:

* History of atrial fibrillation (AF), AF on 12-lead ECG, or any AF of any duration during heart-rhythm monitoring prior to randomization.
* Clear indication for treatment-dose anticoagulant therapy, such as venous thromboembolism or a mechanical heart valve.
* Need for antiplatelet agent, such as aspirin or clopidogrel
* History of spontaneous intracranial hemorrhage.
* Chronic kidney disease with serum creatinine ≥2.5 mg/dL.For Canadian sites only, estimated creatinine clearance (eCrCl) <15 mL/min is also an exclusion criterion.
* Active hepatitis or hepatic insufficiency with Child-Pugh score B or C.
* Clinically significant bleeding diathesis.
* Unresolved anemia (hemoglobin <9 g/dL) or thrombocytopenia (<100 x 10E9/L).
* Clinically significant gastrointestinal bleeding within the past year (e.g., not due to external hemorrhoids).
* At risk for pregnancy: premenopausal or postmenopausal woman within 12 months of last menses without a negative pregnancy test or not committing to adequate birth control, which includes an oral contraceptive, two methods of barrier birth control such as condom with or without spermicidal lubricant + diaphragm, or abstinence.
* Known allergy or intolerance to aspirin or apixaban.
* Concomitant participation in another clinical trial involving a drug or acute stroke intervention.
* Considered by the investigator to have a condition that precludes follow-up or safe participation in the trial.
* Inability of either participant or surrogate to provide written, informed consent for trial participation.

To be eligible for randomization, consented participants must meet criteria for atrial cardiopathy in addition to the inclusion/exclusion criteria above.

Atrial cardiopathy is defined as ≥1 of the following:

* PTFV1 >5,000 μV*ms on 12-lead ECG (ECG criterion).
* Serum NT-proBNP >250 pg/mL (NT-proBNP criterion).
* Left atrial diameter index ≥3 cm/m2 on echocardiogram (i.e., severe left atrial enlargement) (ECHO criterion)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randolph S Marshall, MD, Principal Investigator — Columbia University
Locations (177):
- United States (165):
  - University of Alabama, Birmingham, Alabama
  - University of South Alabama University Hospital, Mobile, Alabama
  - Chandler Regional Medical Center Chandler, AZ, Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Mercy San Juan Medical Center (Dignity Health), Carmichael, California
  - Eden Medical Center, Castro Valley, California
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Fountain Valley Regional Hospital and Medical Center, Fountain Valley, California
  - Community Regional Medical Center, Fresno, California
  - UCSD Health La Jolla, La Jolla, California
  - Sharp Grossmont Hospital, La Mesa, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Los Alamitos Medical Center, Los Alamitos, California
  - Kaiser Permanente, Los Angeles, California
  - Keck Hospital Of USC, Los Angeles, California
  - Los Angeles County- USC Medical Center, Los Angeles, California
  - VA Greater Los Angeles - West LA VA Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Sutter Medical Center, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Scripps Mercy, San Diego, California
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - Kaiser Permanent San Diego Medical Center, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - San Francisco General, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Good Samaritan, San Jose, California
  - Stanford University Medical Center, Stanford, California
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Medical Center, Grand Junction, Colorado
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Med-star Georgetown Univ., Washington D.C., District of Columbia
  - Medstar Washington, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UF Health Shands, Gainesville, Florida
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Jackson Memorial, Miami, Florida
  - Univ. Miami Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Intercoastal Medical Group - Hyde Park, Sarasota, Florida
  - Tampa General, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Grady Memorial, Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Southern Illinois University Memorial Medical Center, Springfield, Illinois
  - St. John's Hospital (Prairie Research), Springfield, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Multi-Specialty - Methodist Plaza/Unity Point, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical, Boston, Massachusetts
  - Brigham & Womens Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - U Mass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Detroit Receiving Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - Mercy Health St. Mary's, Grand Rapids, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - McLaren Macomb, Mount Clemens, MI, Mount Clemens, Michigan
  - McLaren Northern Michigan, Petoskey, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County, Minneapolis, Minnesota
  - Univ. of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital, St. Paul, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Cox Medical Center South, Springfield, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - CHI Health Immanuel, Omaha, Nebraska
  - University of Nebraska, Omaha, Nebraska
  - Cooper University Hospital,, Camden, New Jersey
  - Robert Wood Johnson, New Brunswick, New Jersey
  - Capital Health Medical Center Hopewell, Pennington, New Jersey
  - Univ. New Mexico, Albuquerque, New Mexico
  - Kings County Hospital, Brooklyn, New York
  - New York Presbyterian - Brooklyn Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Mount Sinai Beth Israel Brooklyn, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, Ohio
  - UH Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner, Columbus, Ohio
  - Ohio Health Riverside - Riverside Methodist Hospital, Columbus, Ohio
  - Miami Valley Hospita, Dayton, Ohio
  - Mercy St Vincent Medical Center, Toledo, Ohio
  - OU Medical Center Oklahoma, Oklahoma City, Oklahoma
  - Legacy Emanuel, Portland, Oregon
  - Oregon Health and Sciences, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital (formerly Palmetto Health), Columbia, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Valley Bapist, Harlingen, Texas
  - Baylor College College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Univ of Texas Health Science Center San Antonio, San Antonio, Texas
  - Scott & White Memorial Hospital - Temple, Temple, Texas
  - Memorial Hermann The Woodlands Hospital, The Woodlands, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Univ of Utah, Salt Lake City, Utah
  - George E Whalen VA, Salt Lake City, Utah
  - UVA Medical Center, Charlottesville, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - Providence St. Peter Hospital, Olympia, Washington
  - Harborview Medical Center, Seattle, Washington
  - Puget Sound VA, Seattle, Washington
  - Swedish Medical Center - Cherry Hill Campus, Seattle, Washington
  - WVU Healthcare Ruby Memorial, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (12):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Neurologic Research Center, Lethbridge, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Brandon Regional Health Center, Brandon, Manitoba
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Center, London, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Enfant-Jesus Hospital, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
To share individual participant data (IPD) of baseline characteristics, follow up, outcomes, etc. based on NIH/NINDS requirements.
Supporting Information: Study Protocol
Time Frame: As per NIH/NINDS requirements.
Access Criteria: All items required by NIH/NINDS will be publicly shared.

REFERENCES:
- [Background] Kamel H, Okin PM, Elkind MS, Iadecola C. Atrial Fibrillation and Mechanisms of Stroke: Time for a New Model. Stroke. 2016 Mar;47(3):895-900. doi: 10.1161/STROKEAHA.115.012004. Epub 2016 Jan 19. No abstract available. PMID 26786114
- [Background] Yaghi S, Kamel H, Elkind MS. Potential new uses of non-vitamin K antagonist oral anticoagulants to treat and prevent stroke. Neurology. 2015 Sep 22;85(12):1078-84. doi: 10.1212/WNL.0000000000001817. Epub 2015 Jul 17. PMID 26187229
- [Background] Kamel H, Okin PM, Longstreth WT Jr, Elkind MS, Soliman EZ. Atrial cardiopathy: a broadened concept of left atrial thromboembolism beyond atrial fibrillation. Future Cardiol. 2015 May;11(3):323-31. doi: 10.2217/fca.15.22. PMID 26021638
- [Background] Yaghi S, Moon YP, Mora-McLaughlin C, Willey JZ, Cheung K, Di Tullio MR, Homma S, Kamel H, Sacco RL, Elkind MS. Left atrial enlargement and stroke recurrence: the Northern Manhattan Stroke Study. Stroke. 2015 Jun;46(6):1488-93. doi: 10.1161/STROKEAHA.115.008711. Epub 2015 Apr 23. PMID 25908460
- [Background] Longstreth WT Jr, Kronmal RA, Thompson JL, Christenson RH, Levine SR, Gross R, Brey RL, Buchsbaum R, Elkind MS, Tirschwell DL, Seliger SL, Mohr JP, deFilippi CR. Amino terminal pro-B-type natriuretic peptide, secondary stroke prevention, and choice of antithrombotic therapy. Stroke. 2013 Mar;44(3):714-9. doi: 10.1161/STROKEAHA.112.675942. Epub 2013 Jan 22. PMID 23339958
- [Derived] Marshall RS, Lal BK, Edwards LJ, Huston J, Meschia JF, Brott TG, Howard G, Mena-Hurtado CI, Heck D, Sangha N, Lanzino G, Kashyap VS, Aronow HD, Sharafuddin M, Rai P, Jumani S, Voeks JH, Zhang Y, Slane KJ, Lazar RM, Liebeskind DS; CREST-H investigators. Relationship Between of Degree of Stenosis and Time-To-Peak Delay in High Grade Asymptomatic Carotid Artery Disease. Stroke. 2026 Jan 29. doi: 10.1161/STROKEAHA.125.054149. Online ahead of print. PMID 41608800
- [Derived] Lazar RM, Howard G, Brewer MT, Cassarly C, Pauls Q, Kemp S, Tirschwell DL, Sheth KN, Wintermark M, Kamel H, Longstreth WT Jr, Elkind MSV, Broderick JP, Lansberg MG. Apixaban Versus Aspirin to Reduce Cognitive Decline After Cryptogenic Stroke and Atrial Cardiopathy: ARCADIA-Cognition Study. J Am Heart Assoc. 2025 Sep 16;14(18):e042147. doi: 10.1161/JAHA.125.042147. Epub 2025 Aug 22. PMID 40847528
- [Derived] Elias A, Teraoka JT, Soliman EZ, Elkind MSV, Kamel H, Kronmal RA, Longstreth WT Jr, Tirschwell DL, Di Tullio MR, Marcus GM. Premature Atrial Contractions as a Marker of Atrial Cardiopathy: A Revised Analysis of the ARCADIA Randomized Trial. J Cardiovasc Electrophysiol. 2025 Jul;36(7):1487-1493. doi: 10.1111/jce.16629. Epub 2025 Apr 28. PMID 40294164
- [Derived] Navi BB, Elkind MSV, Zhang C, Tirschwell DL, Kronmal RA, Elm J, Broderick JP, Gladstone DJ, Beyeler M, Kamel H, Longstreth WT Jr. History of Cancer and Atrial Cardiopathy: A Secondary Analysis of the ARCADIA Clinical Trial. J Am Heart Assoc. 2025 May 6;14(9):e040543. doi: 10.1161/JAHA.124.040543. Epub 2025 Apr 23. PMID 40265582
- [Derived] Lansberg MG, Wintermark M, Chen H, Howard G, Cassarly C, Pauls Q, Kemp S, Harris TL, Krishnaiah B, Stanton RJ, Lyerly MJ, Miller BR, Smith EE, Tirschwell DL, Sheth KN, Kamel H, Longstreth WT Jr, Elkind MSV, Broderick JP, Lazar RM. Apixaban to Prevent Covert Infarcts After Cryptogenic Stroke in Patients With Atrial Cardiopathy: A Secondary Analysis of the ARCADIA Randomized Clinical Trial. JAMA Neurol. 2025 Mar 1;82(3):220-227. doi: 10.1001/jamaneurol.2024.4838. PMID 39869342
- [Derived] Navi BB, Zhang C, Miller BR, Pawar A, Cushman M, Kasner SE, Tirschwell D, Longstreth WT, Kronmal R, Elm J, Zweifler RM, Tarsia J, Broderick JP, Gladstone DJ, Beyeler M, Kamel H, Elkind MSV, Streib C. Diagnosis of Incident Cancer After Cryptogenic Stroke: An Exploratory Analysis of the ARCADIA Randomized Trial. Neurology. 2024 Nov 26;103(10):e210027. doi: 10.1212/WNL.0000000000210027. Epub 2024 Oct 31. PMID 39481070
- [Derived] Navi BB, Zhang C, Miller B, Cushman M, Kasner SE, Elkind MSV, Tirschwell DL, Longstreth WT Jr, Kronmal RA, Beyeler M, Elm J, Zweifler RM, Tarsia J, Cereda CW, Bianco G, Costamagna G, Michel P, Broderick JP, Gladstone DJ, Kamel H, Streib C. Apixaban vs Aspirin in Patients With Cancer and Cryptogenic Stroke: A Post Hoc Analysis of the ARCADIA Randomized Clinical Trial. JAMA Neurol. 2024 Sep 1;81(9):958-965. doi: 10.1001/jamaneurol.2024.2404. PMID 39133474
- [Derived] Kamel H, Longstreth WT Jr, Tirschwell DL, Kronmal RA, Marshall RS, Broderick JP, Aragon Garcia R, Plummer P, Sabagha N, Pauls Q, Cassarly C, Dillon CR, Di Tullio MR, Hod EA, Soliman EZ, Gladstone DJ, Healey JS, Sharma M, Chaturvedi S, Janis LS, Krishnaiah B, Nahab F, Kasner SE, Stanton RJ, Kleindorfer DO, Starr M, Winder TR, Clark WM, Miller BR, Elkind MSV; ARCADIA Investigators. Apixaban to Prevent Recurrence After Cryptogenic Stroke in Patients With Atrial Cardiopathy: The ARCADIA Randomized Clinical Trial. JAMA. 2024 Feb 20;331(7):573-581. doi: 10.1001/jama.2023.27188. PMID 38324415
- See also: NIH/NINDS StrokeNet Prevention trials website — https://www.nihstrokenet.org/trials/arcadia/home
- See also: ARCADIA Trial Video — https://youtu.be/YIneZ4n-xXE

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 37,443 potential participants screened, 2,730 were consented by 174 sites into the trial to undergo further criteria review and determine eligibility for randomization by criterion. Once a subject reached eligibility criteria for at least one of the three trial markers, they were approached for randomization. In the end, the study randomized 1,015 subjects at 141 sites (507 in apixaban arm & 508 in aspirin arm).
Pre-assignment Details: 2,730 subjects were consented, then 3 biomarkers were obtained and reviewed for randomization eligibility. 1,015 out of 2,730 were eligible and randomized into the study.
Groups:
- Active Agent: Apixaban: Patients with a recent embolic stroke of undetermined source (ESUS) and evidence of atrial cardiopathy will receive Apixaban
  Apixaban: 5 mg by mouth twice daily (2.5 mg for subjects meeting standard criteria for an adjusted dose) and aspirin placebo once daily.
- Active Control: Aspirin: Patients with a recent embolic stroke of undetermined source (ESUS) and evidence of atrial cardiopathy will receive Aspirin
  Aspirin: Aspirin 81 mg by mouth once daily and apixaban placebo twice daily.
Period: Overall Study
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin
Started | 507 | 508
Completed | 416 | 421
Not Completed | 91 | 87
Not completed — Death | 28 | 23
Not completed — Lost to Follow-up | 10 | 15
Not completed — Withdrawal by Subject | 49 | 48
Not completed — Other as reported in analysis | 4 | 1

BASELINE CHARACTERISTICS:
Population: The initial randomization goal was 1,100 participants but the trial was stopped by the DSMB for futility without any safety concerns at 1,015 randomizations.
Groups:
- Active Agent: Apixaban: Patients with a recent embolic stroke of undetermined source (ESUS) and evidence of atrial cardiopathy will receive Apixaban
  Apixaban: 5 mg by mouth twice daily (2.5 mg for subjects meeting standard criteria for an adjusted dose) and an aspirin placebo once daily.
- Active Control: Aspirin: Patients with a recent embolic stroke of undetermined source (ESUS) and evidence of atrial cardiopathy will receive Aspirin
  Aspirin: Aspirin 81 mg by mouth once daily and an apixaban placebo twice daily.
- Total: Total of all reporting groups
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin | Total
Number analyzed (Participants) | 507 | 508 | 1015
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 202 | 179 | 381
  >=65 years | 305 | 329 | 634
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (10.8) | 68.2 (11.0) | 68.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 279 | 551
  Male | 235 | 229 | 464
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: There were some participants that did not provide this information.
  Participants
    number analyzed (Participants) | 505 | 505 | 1010
    Hispanic or Latino | 43 | 39 | 82
    Not Hispanic or Latino | 462 | 466 | 928
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 107 | 107 | 214
  White | 381 | 379 | 760
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 16 | 32
  United States | 491 | 492 | 983
Weight (kg) [Mean (Standard Deviation); unit: kg] — Population: Not all randomized subjects had weight measurement entered.
  kg
    number analyzed (Participants) | 507 | 506 | 1013
    (all) | 85.1 (20.1) | 84.5 (20.2) | 84.8 (20.2)
CHA2DS2-VASc Score [Mean (Standard Deviation); unit: points in a score system] — The CHA₂DS₂-VASc was developed to be more inclusive of common stroke risk factors/modifiers. Score range is from 0 to 9. Higher score indicates higher risk.
  points in a score system | 4.7 (1.3) | 4.7 (1.3) | 4.7 (1.3)
NIH Stroke Scale [Median (Full Range); unit: score on a scale] — The NIHSS quantifies stroke severity. Score range is from 0 to 42. Higher score shows a more severe stroke. Population: The admission NIHSS was not entered on all randomized subjects.
  score on a scale
    number analyzed (Participants) | 504 | 506 | 1010
    (all) | 1 [0 to 3] | 1 [0 to 3] | 1 [0 to 3]
Atrial Cardiopathy Biomarker - NTproBNP (pg/mL) [Median (Full Range); unit: pg/mL] — NT-proBNP is typically used to determine if certain proteins are increased indicating heart failure. Population: Subjects were eligible for randomization based on at least one biomarker and some did not have all of the three biomarkers measured/entered.
  pg/mL
    number analyzed (Participants) | 502 | 496 | 998
    (all) | 288 [87 to 535] | 318 [130 to 551] | 303 [107 to 547]
Atrial Cardiopathy Biomarker - P-wave terminal force in lead V1 (µV*ms) [Mean (Standard Deviation); unit: µV*ms] — Population: Subjects were eligible for randomization based on at least one biomarker and some did not have all of the three biomarkers measured/entered.
  µV*ms
    number analyzed (Participants) | 501 | 503 | 1004
    (all) | 4,716 (2,515) | 4,766 (2,920) | 4,741 (2,724)
Atrial Cardiopathy Biomarker - Left atrial diameter index (cm/m2; site reported) [Mean (Standard Deviation); unit: cm/m2] — Population: Subjects were eligible for randomization based on at least one biomarker and some did not have all of the three biomarkers measured/entered.
  cm/m2
    number analyzed (Participants) | 406 | 412 | 818
    (all) | 1.9 (0.5) | 1.9 (0.5) | 1.9 (0.5)
Medical Comorbidities - Hypertension [Count of Participants; unit: Participants] | 396 | 388 | 784
Medical Comorbidities - Prior or Current Tobacco Use [Count of Participants; unit: Participants] | 230 | 200 | 430
Medical Comorbidities - Diabetes mellitus [Count of Participants; unit: Participants] | 156 | 159 | 315
Medical Comorbidities - Prior stroke or TIA [Count of Participants; unit: Participants] | 97 | 100 | 197
Medical Comorbidities - Ischemic Heart Disease [Count of Participants; unit: Participants] | 58 | 46 | 104
Medical Comorbidities - Heart Failure [Count of Participants; unit: Participants] | 36 | 35 | 71
Medical Comorbidities - Peripheral Arterial Disease [Count of Participants; unit: Participants] | 12 | 7 | 19
Days from index stroke to randomization [Median (Inter-Quartile Range); unit: days] | 48 [21 to 96] | 53 [23 to 100] | 50 [22 to 97]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Stroke of Any Type
Description: Participants were monitored for up to 5 years of study participation. This is the number of participants who had recurrent stroke of any type (ischemic, hemorrhagic, or of unclear type).
Time Frame: Up to 5 years of study participation.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin
Number analyzed (Participants) | 507 | 508
Participants | 40 | 40
Statistical Analysis 1: Comparison: Active Agent: Apixaban vs Active Control: Aspirin; Test type: Superiority; p = 0.99, Log Rank; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.64 to 1.55]

2. Secondary Outcome: Number of Participants With Recurrent Ischemic Stroke or Systemic Embolism
Description: Secondary efficacy outcome A. Participants were monitored for up to 5 years. This is the number of participants who had recurrent ischemic stroke or systemic embolism during the time of observation.
Time Frame: Up to 5 years of study participation.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin
Number analyzed (Participants) | 507 | 508
Participants | 37 | 40
Statistical Analysis 1: Comparison: Active Agent: Apixaban vs Active Control: Aspirin; Test type: Superiority; p = 0.72, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.59 to 1.44]

3. Secondary Outcome: Number of Participants With Recurrent Stroke of Any Type or Death From Any Cause
Description: Secondary efficacy outcome B. Participants were monitored for up to 5 years. This is the number of participants who had recurrent stroke of any type or death from any cause during the observation time.
Time Frame: Up to 5 years of study participation.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin
Number analyzed (Participants) | 507 | 508
Participants | 67 | 62
Statistical Analysis 1: Comparison: Active Agent: Apixaban vs Active Control: Aspirin; Test type: Superiority; p = 0.67, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.76 to 1.52]

4. Secondary Outcome: Number of Participants With Symptomatic Intracranial Hemorrhage (Including Symptomatic Hemorrhagic Transformation of an Ischemic Stroke)
Description: Primary safety outcome A. This is the number of participants who had symptomatic intracranial hemorrhage from any cause during the time of observation. Symptomatic intracranial hemorrhage includes symptomatic hemorrhagic transformation of ischemic stroke, which required new symptoms or signs adjudicated as being due to the hemorrhagic transformation or a patient whose initial imaging was judged to include hemorrhagic transformation of an ischemic stroke.
Time Frame: Through 30 days after permanent discontinuation of the study drug, a duration of up to 5 years for each participant.
Population: The safety sample includes all participants who are randomized and receive at least one dose of study medication.
  The safety sample will include all safety outcomes from randomization until 30 days after permanent discontinuation of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin
Number analyzed (Participants) | 482 | 493
Participants | 0 | 7
Statistical Analysis 1: Comparison: Active Agent: Apixaban vs Active Control: Aspirin; Test type: Superiority; p = .02, Exact Binomial Test; Difference of annual rate. = -0.011, 95% CI 2-sided [-0.018 to -0.003]

5. Secondary Outcome: Number of Participants With Major Hemorrhage Other Than Intracranial Hemorrhage.
Description: This is the number of participants who had major hemorrhage other than intracranial hemorrhage.
Time Frame: Through 30 days after permanent discontinuation of the study drug, a duration of up to 5 years for each participant.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin
Number analyzed (Participants) | 482 | 493
Participants | 5 | 5
Statistical Analysis 1: Comparison: Active Agent: Apixaban vs Active Control: Aspirin; Test type: Superiority; p = 0.98, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.29 to 3.52]

6. Secondary Outcome: Number of Participant Deaths From Any Cause Number of Participants With All-cause Mortality.
Description: Secondary safety outcome. This is the number of participants who had all-cause mortality during time of observation.
Time Frame: Through 30 days after permanent discontinuation of the study drug, a duration of up to 5 years for each participant.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin
Number analyzed (Participants) | 482 | 493
Participants | 12 | 8
Statistical Analysis 1: Comparison: Active Agent: Apixaban vs Active Control: Aspirin; Test type: Superiority; p = 0.35, Log Rank; Hazard Ratio (HR) = 1.53, 95% CI 2-sided [0.63 to 3.75]

ADVERSE EVENTS:
Time Frame: The adverse event data was collected for up to 5 years of study participation via questionnaires used at every follow-up visit. The all-cause mortalities were reported for all the randomized subjects through the whole follow up period of up to 5 plus the mortalities occurred during the adjudication process for the recurrent stroke (primary outcome) and the mortalities occurred more than 30 days after the study medication permanently stopped, up to 61 months.
Description: SAE definition excludes these hospitalizations: to Emergency room/other hospital department <24 hours, not resulting in admission (unless medically important/life-threatening); elective surgery planned prior to study entry; planned medical/surgical procedure; routine health assessment requiring medical/surgical admission other than to remedy ill health/planned prior to study entry; for another life circumstance w/o bearing on health status/requires no medical/surgical intervention.
Arm/Group | Active Agent: Apixaban | Active Control: Aspirin
All-Cause Mortality (participants affected / at risk) | 32/507 | 24/508
Serious Adverse Events (participants affected / at risk) | 355/507 | 388/508
Other Adverse Events (participants affected / at risk) | 99/507 | 91/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Agent: Apixaban (N=507) | Active Control: Aspirin (N=508)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 7 (7) | 6 (6)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 74 (74) | 77 (77)
Atrial flutter (Cardiac disorders) | 1 (1) | 4 (4)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 7 (8) | 8 (9)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 5 (5) | 5 (5)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 3 (3) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 2 (4)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 5 (5)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 4 (4)
Death (General disorders) | 5 (5) | 2 (2)
Necrosis (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 12 (14) | 7 (7)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (3) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 2 (2)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 13 (13) | 11 (12)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 7 (8)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2) | 0 (0)
Basal ganglia stroke (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 8 (8) | 6 (7)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 3 (3)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 29 (29) | 33 (33)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (2) | 0 (0)
Quadriplegia (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 10 (11) | 10 (10)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 6 (7)
Transient ischaemic attack (Nervous system disorders) | 5 (5) | 7 (7)
Vertebral artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 1 (1)
Uncoded (General disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 9 (10) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (5) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 6 (7)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Agent: Apixaban (N=507) | Active Control: Aspirin (N=508)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 33 (34) | 38 (38)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 7 (7)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Coronavirus test positive (Investigations) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Polymerase chain reaction positive (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 4 (4)
Haematuria (Renal and urinary disorders) | 5 (5) | 4 (4)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 2 (3)
Haemorrhage (Vascular disorders) | 4 (4) | 5 (6)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03192215/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03192215/SAP_001.pdf